CLINICAL TRIAL: NCT01949610
Title: Absorption, Metabolism, and Excretion of 14C-JNJ26489112 After a Single Oral Dose in Healthy Male Subjects
Brief Title: A Study to Evaluate Absorption, Metabolism, and Excretion of 14C-JNJ26489112 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016981; 26489112MDD1001 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; JNJ26489112; 14C-JNJ26489112; Absorption; Metabolism; Excretion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 14C-JNJ26489112 (Experimental)
  Interventions: Drug: 14C-JNJ26489112

INTERVENTIONS:
Drug: 14C-JNJ26489112 — Participants will receive single dose of oral suspension of 1000 mg (10 mL) of 14C-JNJ26489112 on Day 1.

SUMMARY:
The purpose of this study is to evaluate the absorption, the metabolic pathways (a series of metabolic reactions) and the excretion of JNJ26489112 in healthy male adult participants after administration of a single oral dose of 1000 mg of 14C-JNJ26489112.

DETAILED DESCRIPTION:
This is a single-dose, 1-arm (group), open-label study (all people know the identity of the intervention) in healthy adult male participants. On Day 1, after completing a 10-hour overnight fast, participants will receive a single oral dose of 14C-JNJ-26489112 1,000 mg as a 10-mL suspension. Participants will be recruited in 2 cohorts. The 6 participants in the first cohort were dosed in error with doses less than 1000 mg. So, an additional cohort of 4 participants will be enrolled to receive a single oral dose of 1000 mg 14C-JNJ 26489112. Total 10 participants will receive the study medication. Safety will be assessed by monitoring vital signs, physical examinations, electrocardiograms, and clinical laboratory tests throughout the study. The total duration of the study for each participant will be approximately 5 weeks (including up to 3 weeks for screening and 11 to 15 days of study) or up to 1 additional week for participants who excrete 14C-JNJ26489112 more slowly.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study, are willing to participate in the study, and are willing to adhere to the prohibitions and restrictions specified in the protocol
* Had consistent bowel movement habit (approximately once per day) within 30 days before dosing
* Blood pressure (after the participant is supine for 5 minutes) is between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic
* A 12-lead electrocardiogram consistent with normal cardiac conduction and function

Exclusion Criteria:

* Exposure to radiation for professional or medical reasons with the exception of up to 2 standard diagnostic radiographs (eg, dental X-rays, plain chest X-ray) or participation in any investigational study involving radioactivity within 1 year before study drug administration on Day 1
* History of or current clinically significant medical illness including cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or at admission to the study center
* Clinically significant abnormal physical examination, vital signs or 12-lead electrocardiogram at screening or at admission to the study center
* Clinically significant ocular deficits, including retinal disorders

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of 14C-JNJ-26489112 in plasma | 240 hours
Mass balance after an oral dose of 14C-JNJ-26489112 as generated from recovery of total radioactivity excreted in urine and feces | 240 hours
Routes of 14C-JNJ-26489112 elimination measured through total radioactivity concentrations in urine and feces | 240 hours
Whole blood and plasma partitioning of total radioactivity through measurement of total radioactivity levels in blood | 240 hours
Identification of major metabolites in plasma, urine, and feces | 240 hours

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to Day 15
Number of participants with a suicide-related outcome | Screening (Days -21 to -1), Day 2 and end-of-study (Day 15)
  Suicide related outcome measures will be assessed by using Columbia-Suicide Severity Rating Scale (C-SSRS). By using the C-SSRS, potential suicide-related events will be categorized using the codes defined by the Columbia Classification Algorithm of Suicide Assessment from Code 0: no event that can be assessed based on the C-SSRS to Code 9: not enough information, nonfatal. The 4 suicide-related outcomes of interest are the following: suicidal ideation (Code 4), suicidal behavior (Codes 1 to 3), suicidal behavior or ideation (Codes 1 to 4), and possible suicidal behavior or ideation (Codes 1 to 6 and 9).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Merksem, Belgium